CLINICAL TRIAL: NCT03837730
Title: Activity and Expression of Plasma Arginase in Patients With Severe Sepsis or Septic Shock as Prognostic Value
Brief Title: Citrulline and Arginase Activity in Severe Sepsis and Septic Shock
Acronym: CARS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2018/353
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Intensive Care Units; Infection; Biomarkers; Sepsis; Septic Shock
Keywords: ICU, sepsis, septic shok, arginase, citrulline
MeSH Terms: conditions — Infections; Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample at ICU admission, day 3 and day 7 biomarkers analysis: arginase activity, citrulline and IFABP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sepsis is an acute pathology defined as an inappropriate response of the host to infection, resulting in the onset of organ failure (Quick SOFA ≥2, or SOFA ≥2). Septic shock is a sepsis associated with an elevation of lactate ≥ 2 mmol / l and an arterial hypotension requiring vasoactive drugs. Several studies highlighted that sepsis is associated with a plasma L-arginine deficiency. This deficiency induces a lower availability of L-arginine for multiple metabolic pathways including those involved in the synthesis of nitric oxide (NO) in the vascular endothelium via NO synthase. NO is the main endogenous vasodilator mediator, a lower synthesis induces a vascular and endothelial dysfunction that can promote the occurrence of an organic dysfunction during sepsis. Decrease in available NO was confirmed in patients with sepsis and appears correlated with severity.

L-arginine deficiency can have multiple origins:

* L-arginine deficiency resulting from a decrease in endogenous production from citrulline synthesized by the enterocytes. Such enterocyte dysfunction has been confirmed in patients with sepsis and is characterized biologically by elevated plasma levels of I-FABP (intestinal fatty acid binding protein - enterocyte-specific protein, cytolysis marker) and lower than that of citrulline (hypocitrullinemia, marker of lower activity).
* L-arginine deficiency may also result from a catabolism increase via arginase activity increased. This ubiquitous enzyme, having 2 isoforms (Arg1 and Arg2), allows the synthesis of urea and ornithine from L-arginine. An increase in arginase activity would decrease the available reserves of L-arginine for NO synthesis.

The objectives of this work is to evaluate, in patients with severe sepsis or septic shock, the prognostic value of the plasma arginase activity and the plasma expression of 2 isoforms Arg1 and Arg2, their kinetics, and the link between activity / expression of arginase and enterocyte dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Patient admitted to ICU
* Diagnosis, suspected or confirmed, of severe sepsis or septic shock
* Expected ICU stay of at least 2 days
* Affiliation to a social security system or recipient of a such system
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Chronic intestinal pathology
* Chronic renal failure defined by creatinine clearance <50 ml / min / 1.73m2 (CKD-EPI)
* Severe hepatic insufficiency (Child-Pugh stage C score)
* Legal incapacity or limited legal capacity
* Subject unlikely to cooperate with the study and / or weak cooperation anticipated by the investigator
* Patient within the exclusion period of another study or planned by the "national file of volunteers"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to the ICU for severe sepsis or septic shock
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
prognostic value of plasma arginase activity and expression at ICU admission in patients with severe sepsis or septic shock | 28 days
  activity / expression of plasma arginase at ICU admission and 28-day mortality rate from admission to intensive care

SECONDARY OUTCOMES:
activity / expression kinetic of plasma arginase | during the first 7 days of ICU admission
  3 points kinetic : admission, day 3 and day 7
prognostic value of enterocyte damage | 28 days
  at ICU admission and 28-day mortality rate from admission to intensive care

CONTACTS AND LOCATIONS:
Overall Officials: Gaël PITON, MD, Principal Investigator — CHU DE BESANCON
Locations (1):
- CHU de BESANCON, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided